CLINICAL TRIAL: NCT03836508
Title: Effect of Dialysis Membranes on Inflammatory and Immune Processes in Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nuri Baris Hasbal, Principal Investigator, MD, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 1909
Record Dates: First submitted 2019-01-20; First posted 2019-02-11 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Kidney Failure; Renal Insufficiency, Chronic; Dialysis Related Complication
MeSH Terms: conditions — Renal Insufficiency; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medium cut-off (Active Comparator): Medium cut-off dialyzers will be used in this group containing 26 randomized patients for three months. At the end of the third month with crossover, this groups of patients will start using high-flux dialyzers.
  Interventions: Device: Medium cut-off; Device: High-Flux
- High-flux (Active Comparator): High-flux dialyzers will be used in this group containing 26 randomized patients for three months. At the end of the third month with crossover, this groups of patients will start using medium cut-off dialyzers.
  Interventions: Device: Medium cut-off; Device: High-Flux

INTERVENTIONS:
Device: Medium cut-off — All the dialysis sessions in this arm will be performed with the medium cut-off membrane (MCO) manufactured by Baxter International Corp. membrane for three months. This membrane will exclusively be used in hemodialysis. After third month, all patients will be switched to high-flux membrane manufactured by Fresenius.
  Modalities of hemodialysis : Blood flow: 300-400 mL/min; Dialysate flow: 500-800 mL/min
Device: High-Flux — All the dialysis sessions in this arm will be performed with the high-flux membrane manufactured by Fresenius for three months. This membrane will exclusively be used in hemodialysis. After third month, all patients will be switched to MCO manufactured by Baxter International Corp.
  Modalities of hemodialysis : Blood flow: 300-400 mL/min; Dialysate flow: 500-800 mL/min

SUMMARY:
Double blinded, randomized controlled trial evaluating medium cut-off dialyzer compared to high flux dialyzer in ironic hemodialysis patients over a 6 months period with 3 months crossovers.

ELIGIBILITY:
Inclusion Criteria:

* patients who are older than 18 years and younger than 65 years
* patient with end-stage renal disease, hemodialysis more than 6 months
* patients under hemodialysis with high-flux dialyzer more than 3 months
* patients willing to participate after given fair and clear information about study

Exclusion Criteria:

* patients living with Hepatitis B or C,
* patients with malignancy
* patients under immunosuppressive treatment
* patients with autoimmune diseases such as systemic lupus erythematosus, etc.
* patients with active infections
* patients planned to have a kidney transplantation in 6 months
* patients having vascular access problems
* patients planned to transfer to another center

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Comparison of pre and post-dialysis of Interleukin (IL) 17-A | 3 months
  Comparison of pre and post-dialysis of IL-17A

SECONDARY OUTCOMES:
Comparison of pre and post-dialysis of IL-10 | 3 months
  Comparison of pre and post-dialysis of IL-10
Comparison of pre and post-dialysis of Interferon (IFN) gama | 3 months
  Comparison of pre and post-dialysis of IFN gama
Comparison of pre and post-dialysis necrosis factor (TNF) alpha | 3 months
  Comparison of pre and post-dialysis of TNF alpha
Comparison of pre and post-dialysis of IL-4 | 3 months
  Comparison of pre and post-dialysis of IL-4
Comparison of pre and post-dialysis of Urea | 3 months
  Comparison of pre and post-dialysis of Urea
Comparison of pre and post-dialysis of creatinine | 3 months
  Comparison of pre and post-dialysis of creatinine
Comparison of pre and post-dialysis of beta2 microglobulin | 3 months
  Comparison of pre and post-dialysis of beta2 microglobulin
Comparison of pre and post-dialysis of free light chain kappa | 3 months
  Comparison of pre and post-dialysis of free light chain kappa
Comparison of pre and post-dialysis of free light chain lambda | 3 months
  Comparison of pre and post-dialysis of free light chain lambda
Comparison of pre and post-dialysis of myoglobulin | 3 months
  Comparison of pre and post-dialysis of myoglobulin
Comparison of pre and post-dialysis of fibroblast growth factor (FGF) 23 | 3 months
  Comparison of pre and post-dialysis of FGF 23
Comparison of pre and post-dialysis IL-18 levels | 3 months
  Comparison of pre and post-dialysis IL-18 levels
Comparison of pre and post-dialysis monocyte chemoattractant protein (MCP)-1 levels | 3 months
  Comparison of pre and post-dialysis MCP-1 levels
Comparison of pre and post-dialysis NACHT, LRR and PYD domains-containing protein3 (NLRP3) levels | 3 months
  Comparison of pre and post-dialysis NLRP3 levels
Comparison of pre and post-dialysis regulated on activation, normal T cell expressed and secreted (RANTES) | 3 months
  Comparison of pre and post-dialysis RANTES

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Sevinc, MD, Principal Investigator — Sisli Hamidiye Etfal Training and Research Hospital
Locations (1):
- Sisli Hamidiye Etfal Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-27): https://cdn.clinicaltrials.gov/large-docs/08/NCT03836508/Prot_SAP_000.pdf